CLINICAL TRIAL: NCT02962726
Title: Microbiome Shifts in Adolescent Anorexia Nervosa
Acronym: MaAN
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-093
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia; Depression; Microbiome
MeSH Terms: conditions — Anorexia Nervosa; Anorexia; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: 100 female patients between the age of 12 and 18 years suffering from anorexia nervosa.
- Age matched Controls: 100 females volunteers between the age of 12 and 18 years old without eating disorder.

SUMMARY:
The aim of this study is to evaluate the effect of starvation and recovery in adolescent anorexia nervosa patients in regard to microbiome activity and composition and to elucidate potential connections between weight gain, depression and other comorbidities, further to capture hormone levels and inflammation parameters in a longitudinal design.

DETAILED DESCRIPTION:
Anorexia Nervosa (AN) has the highest mortality of all psychiatric disorders. Large part of all patients the disorder becomes chronical. Until now, no (bio-) markers which allow a prognosis of outcome are known. Recently the function of the intestinal microbiome and its effects on food uptake, immunological processes and barrier malfunctions in the intestine is discussed. Especially the concept of the "leaky gut", an adsorption malfunction of the intestinal wall under starvation for antigens may help to explain the low inflammatory response which is commonly found in Anorexia Nervosa subjects and a connection to higher rate of autoimmune diseases by Anorexia Nervosa. Furthermore the presence and quantity of specific bacteria in the intestine seems to be dependent on patient's sex which would contribute to the gender gap of prevalence for Anorexia Nervosa. Stress induced changes of the HPA-axis which are well documented in Anorexia Nervosa patients and often persist even after weight rehabilitation, play an important part for intestinal wall permeability disorders. In the most often used animal model for AN, the Activity-Based Anorexia (ABA) model which combines nutrition restriction and weight loss with hyper activity, a malfunction in intestinal wall permeability was found. Malnutrition and long lasting dieting have a fast and reproducible impact on the intestinal microbiome. Especially animal derived food seems to support proliferation of pro-inflammatory bacteria. A substantial intestinal dysbiosis (reduced alpha-diversity) was found in AN patients which only partly recovered after weight rehabilitation. Reduction in diversity and composition of the microbiome was significantly associated with severity of depressive symptoms in patient, where severity is an indicator for higher level eating pathologies and poorer prognosis. Aim of this longitudinal study is therefore to investigate to interconnections between fecal microbiome and progression of AN, including associations with stress, inflammatory markers and metabolic markers in blood sera as well as clinical parameters such as severity of depression and eating pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Female patients and volunteers between age 12 and 18 at inclusion.
* Written informed consent by Patient/volunteer and caregiver.
* Volunteers with BMI between 10 and 90 percentile of their age group.
* Volunteers without prior eating or mental disorder.

Exclusion Criteria:

* Psychotic disorder(s)
* Personality disorder(s)
* Alcohol and substance abuse
* Prone to self-harming behaviour
* Primary caregiver insufficient German language skills
* Patient/Volunteers IQ lower 85
* Antibiotic treatment within 4 weeks prior to inclusion

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 100 female patients suffering from anorexia nervosa. 100 female volunteers without eating or mental disorder.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation BMI and Microbiome Variability | 12 month
  Correlation between Body Mass Index and Microbiome Variability.

SECONDARY OUTCOMES:
Bacteria | 12 month
  Qualitative description of bacteria species
Bacteria activity | 12 month
  Quantitative description of Bacterial activity
Inflammatory parameters | 12 month
Depression | 12 month
  Depression assessment Beck's Depression Inventory II

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Seitz, MD, Principal Investigator — University Hospital, Aachen
Locations (1):
- Clinic for Paediatric Psychiatry, Psychosomatic Disorders and Psychotherapy, Aachen, North Rhine Westphali, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herpertz-Dahlmann B. Adolescent eating disorders: update on definitions, symptomatology, epidemiology, and comorbidity. Child Adolesc Psychiatr Clin N Am. 2015 Jan;24(1):177-96. doi: 10.1016/j.chc.2014.08.003. Epub 2014 Oct 7. PMID 25455581
- [Background] Raevuori A, Haukka J, Vaarala O, Suvisaari JM, Gissler M, Grainger M, Linna MS, Suokas JT. The increased risk for autoimmune diseases in patients with eating disorders. PLoS One. 2014 Aug 22;9(8):e104845. doi: 10.1371/journal.pone.0104845. eCollection 2014. PMID 25147950
- [Background] Solmi M, Veronese N, Favaro A, Santonastaso P, Manzato E, Sergi G, Correll CU. Inflammatory cytokines and anorexia nervosa: A meta-analysis of cross-sectional and longitudinal studies. Psychoneuroendocrinology. 2015 Jan;51:237-52. doi: 10.1016/j.psyneuen.2014.09.031. Epub 2014 Oct 8. PMID 25462897
- [Background] Corcos M, Guilbaud O, Paterniti S, Moussa M, Chambry J, Chaouat G, Consoli SM, Jeammet P. Involvement of cytokines in eating disorders: a critical review of the human literature. Psychoneuroendocrinology. 2003 Apr;28(3):229-49. doi: 10.1016/s0306-4530(02)00021-5. PMID 12573293
- [Background] Tennoune N, Legrand R, Ouelaa W, Breton J, Lucas N, Bole-Feysot C, do Rego JC, Dechelotte P, Fetissov SO. Sex-related effects of nutritional supplementation of Escherichia coli: relevance to eating disorders. Nutrition. 2015 Mar;31(3):498-507. doi: 10.1016/j.nut.2014.11.003. Epub 2014 Dec 5. PMID 25701341